CLINICAL TRIAL: NCT07309887
Title: Real-world Characteristics and Risk of Disease Recurrence in Hormone Receptor-positive, HER2-negative Early Breast Cancer: a Multi-center Retrospective Cohort Study in Korea
Brief Title: This Clinical Trial is a Retrospective, Multicenter Cohort Study Evaluating the Real-world Characteristics and Risk of Disease Recurrence in Hormone Receptor-positive, HER2-negative Early Breast Cancer.
Acronym: PRIORITY
Status: Not yet recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Yeon Hee Park, Clinical Professor, Samsung Medical Center
Other Study IDs: 2025-08-005
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Early Breast Cancer
Keywords: Early breast cancer retrospective cohort study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Primary objective: To describe event-free survival (EFS) in patients with stage I-III HR+/HER2- early breast cancer (EBC) who received curative surgery followed by systemic therapy.
* Secondary objectives: Include assessment of relapse-free survival (RFS), distant disease-free survival (DDFS), distant relapse-free survival (DRFS), overall survival (OS), site of distant recurrence, and time-to-next treatment (TTNT), as well as evaluating the association between clinicopathologic/treatment variables and clinical outcomes.
* Key inclusion criteria: Adults (≥18 years) with stage I-III HR+/HER2- invasive breast cancer who underwent curative surgery
* Key exclusion criteria: HR- or HER2+ tumors, de novo stage IV, or lack of curative-intent surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients (female or male) with a histologically confirmed first diagnosis of invasive breast cancer, identified by International Classification of Diseases, 10th Revision (ICD-10) code C50.x, between January 1, 2010, and December 31, 2023.* The date of diagnosis will be based on the initial pathology report or the date reported to the Korea Central Cancer Registry (KCCR).
2. Age 18 years or older at the time of initial diagnosis.
3. Anatomical stage I, II, or III disease at initial diagnosis, staged according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual, using the edition contemporary to the time of diagnosis.
4. Confirmed HR-positive disease, defined as estrogen receptor (ER) and/or progesterone receptor (PR) expression in ≥1% of invasive tumor cells on immunohistochemistry (IHC), or an Allred proportion score of 2 or higher.
5. Confirmed HER2-negative disease, defined as an IHC score of 0 or 1+, or an IHC score of 2+ with a negative in situ hybridization (ISH) result (e.g., fluorescence in situ hybridization or silver in situ hybridization). Patients recorded as HER2-negative without a specific score available will also be included.
6. Documented history of having received definitive (curative-intent) surgery for the primary breast cancer (e.g., breast-conserving surgery or mastectomy).

Exclusion Criteria:

1. Patients (female or male) with a histologically confirmed first diagnosis of invasive breast cancer, identified by International Classification of Diseases, 10th Revision (ICD-10) code C50.x, between January 1, 2010, and December 31, 2023.* The date of diagnosis will be based on the initial pathology report or the date reported to the Korea Central Cancer Registry (KCCR).
2. Age 18 years or older at the time of initial diagnosis.
3. Anatomical stage I, II, or III disease at initial diagnosis, staged according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual, using the edition contemporary to the time of diagnosis.
4. Confirmed HR-positive disease, defined as estrogen receptor (ER) and/or progesterone receptor (PR) expression in ≥1% of invasive tumor cells on immunohistochemistry (IHC), or an Allred proportion score of 2 or higher.
5. Confirmed HER2-negative disease, defined as an IHC score of 0 or 1+, or an IHC score of 2+ with a negative in situ hybridization (ISH) result (e.g., fluorescence in situ hybridization or silver in situ hybridization). Patients recorded as HER2-negative without a specific score available will also be included.
6. Documented history of having received definitive (curative-intent) surgery for the primary breast cancer (e.g., breast-conserving surgery or mastectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Key inclusion criteria: Adults (≥18 years) with stage I-III HR+/HER2- invasive breast cancer who underwent curative surgery Key exclusion criteria: HR- or HER2+ tumors, de novo stage IV, or lack of curative-intent surgery
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EFS (Event Free Survival) | Its temporal window, which spans from 2010 to 2023
  The time from the index date (date of initiation of first systemic therapy or date of curative surgery, whichever occurs first) to the date of the first occurrence of any of the following events: disease progression that precludes the ability to perform definitive surgery (for patients receiving neoadjuvant therapy), invasive local or distant recurrence, the occurrence of a second primary invasive cancer, or death from any cause.

SECONDARY OUTCOMES:
RFS | Its temporal window, which spans from 2010 to 2023
  Time from index date to any recurrence (local/regional/distant) or death from any cause
DDFS | Its temporal window, which spans from 2010 to 2023.
  Time from index date to distant recurrence, second non-breast primary cancer, or death from any cause
DRFS | Its temporal window, which spans from 2010 to 2023
  Time from index date to distant recurrence or death from any cause
OS | Its temporal window, which spans from 2010 to 2023
  Time from index date to death from any cause
Site of initial distant recurrence | Its temporal window, which spans from 2010 to 2023
  The anatomical location(s) of the first documented distant metastatic lesion(s)
TTNT | Its temporal window, which spans from 2010 to 2023
  Time from the initiation of first-line systemic therapy for advanced/metastatic disease to the initiation of a subsequent line of therapy or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided later.